CLINICAL TRIAL: NCT01892878
Title: A Prospective, Single Arm Clinical Trial Evaluating Clinical Outcome and Fusion Results Using the VerteLoc® Facet Fixation Device
Brief Title: Clinical Outcome and Fusion Results Using the VerteLoc® Facet Fixation Device
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: VG Innovations, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VGI-002
Record Dates: First submitted 2013-07-01; First posted 2013-07-08 (Estimated); Last update posted 2018-03-16 (Actual); Status verified 2013-07

CONDITIONS: Spinal Stenosis
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm Study (Other): All patients will receive treatment
  Interventions: Procedure: VerteLoc

INTERVENTIONS:
Procedure: VerteLoc — Single Arm

SUMMARY:
The purpose of this clinical study is to evaluate fusion of the facet joints in a prospective cohort of patients utilizing the VerteLoc facet fixation device in patients receiving lumbar laminectomy (L1-S1), without ancillary stabilization devices such as pedicle and transfacet screws.

DETAILED DESCRIPTION:
Study Design: Non-randomized, prospective, single arm clinical trial

Patient Population and Sample Size: Patients (n=25) from up to 2 clinical site, who have been medically evaluated, found appropriate for, and have agreed to treatment by lumbar decompressive laminectomy and facet fixation, including unilateral and/or bilateral posterolateral fusion according to accepted medical standards.

Objectives:

The primary objective of this study is to:

1. Evaluate the fusion status of facet joints following laminectomy and facet fixation using the VerteLoc system in combination with unilateral and/or bilateral posterolateral fusion.
2. Subject success / Clinical outcome: Evaluate the reduction in baseline VAS back pain score at 2-3 weeks, 3 months, and 12 months.

The secondary objectives of this study are to:

1. Explore the effect of preoperative bone density on facet fusion status;
2. Assess the ease of use of the VerteLoc system;
3. Record operative time using the VerteLoc system;
4. Monitor the occurrence of adverse events related or possibly related to the use of the VerteLoc system;
5. Monitor the occurrence of subsequent surgical intervention at the target level(s).
6. Subject success/Clinical outcome (Assess additional improvement criteria)
7. Evaluate Fusion rate in relations to DEXA value

Inclusion Criteria: Candidates must meet ALL of the following:

1. Have provided consent for research by signing the Institutional Review Board approved Informed Consent;
2. Have given appropriate operative consent for a decompressive lumbar (L1-S1) laminectomy procedure as standard of care;
3. Are skeletally mature, and are at least 18 years of age;
4. If female, are not pregnant;
5. Agree to adhere to post-surgical medically prescribed activity limitations and/or physical rehabilitation.

Exclusion Criteria:

1. Previous surgery at the target or adjacent vertebral levels;
2. More than two intervertebral levels to be treated by the laminectomy procedure;
3. Found to be inappropriate candidates for facet fixation using the VerteLoc system;
4. Require additional and/or other surgical technique and/or approach to the laminectomy at the index level(s), which may in the opinion of the Primary Investigator confound measurement of outcome variables;
5. Has a medical disorder or is receiving medications that would be expected to interfere with osteogeneses,
6. Active malignancy or patient with a history of any malignancy (except non-melanoma skin cancer) with recurrence within 5 years of surgery;
7. Active local or systemic infection or history of local or systemic infection, immune-deficiency, uncontrolled medical conditions, which in the opinion of the Investigator may increase patient risk or confound fusion results;
8. BMI >40% ;
9. History of tobacco smoking within the past 6 months;
10. Has a history of alcoholism, medication or drug abuse, psychosis, is a prisoner, and/or has a personality disorder, poor motivation, emotional or intellectual issues that would likely make the patient unreliable for participation in the study;
11. Are participating in any other clinical trial. Study Duration : 12 months

Study Outcomes:

The primary study outcomes of this study are:

1. Fusion grade at 12 month follow-up using CT scans with a grading system based on:

   1. Complete fusion;
   2. Partial fusion;
   3. No fusion;
2. Subject success / Clinical outcome:

Evaluate the reduction in baseline VAS back pain score at:

1. 2-3 weeks
2. 3 months
3. 12 months.

The secondary outcomes of this study are:

1. Statistical correlation of DEXA scan bone mass density score to CT and radiographic fusion status;
2. Surgeon opinion of "ease of use" utilizing the VerteLoc system (0-10);
3. Operative time (minutes) from surgical access to completion of device placement
4. Occurrence and prevalence of adverse events related or possibly related to the use of the VerteLoc System;
5. Occurrence of subsequent surgical intervention at the target level(s).

Study Assessments

* Intraoperative: Post-placement radiograph;
* 12 months: A/P and lateral flexion and extension lumbar radiograph and lumbar CT scan.

Statistical Analysis

• Student t-tests

ELIGIBILITY:
Inclusion Criteria:

1. Have provided consent for research by signing the Institutional Review Board approved Informed Consent;
2. Have given appropriate operative consent for a decompressive lumbar (L1-S1) laminectomy procedure as standard of care;
3. Are skeletally mature, and are at least 18 years of age;
4. If female, are not pregnant;
5. Agree to adhere to post-surgical medically prescribed activity limitations and/or physical rehabilitation.

Exclusion Criteria:

1. Previous surgery at the target or adjacent vertebral levels;
2. More than two intervertebral levels to be treated by the laminectomy procedure;
3. Found to be inappropriate candidates for facet fixation using the VerteLoc system;
4. Require additional and/or other surgical technique and/or approach to the laminectomy at the index level(s), which may in the opinion of the Primary Investigator confound measurement of outcome variables;
5. Has a medical disorder or is receiving medications that would be expected to interfere with osteogeneses,
6. Active malignancy or patient with a history of any malignancy (except non-melanoma skin cancer) with recurrence within 5 years of surgery;
7. Active local or systemic infection or history of local or systemic infection, immune-deficiency, uncontrolled medical conditions, which in the opinion of the Investigator may increase patient risk or confound fusion results;
8. BMI >40% ;
9. History of tobacco smoking within the past 6 months;
10. Has a history of alcoholism, medication or drug abuse, psychosis, is a prisoner, and/or has a personality disorder, poor motivation, emotional or intellectual issues that would likely make the patient unreliable for participation in the study;
11. Are participating in any other clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-07; Primary Completion 2015-07 (Estimated); Study Completion 2016-01-01 (Estimated)

PRIMARY OUTCOMES:
Fusion grade at 12 month follow-up using CT scans | 12 months
  Fusion grade at 12 month follow-up using CT scans with a grading system based on:
  1. Complete fusion;
  2. Partial fusion;
  3. No fusion;

SECONDARY OUTCOMES:
Subject success / Clinical outcome | 2-3 weeks, 3 months and 12 months
  Subject success / Clinical outcome:
  Evaluate the reduction in baseline VAS back pain score.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Guyot, MD, Principal Investigator — Ascension Health
Locations (1):
- Genesys Regional Medical Center, Grand Blanc, Michigan, United States